CLINICAL TRIAL: NCT05053087
Title: A Three-Arm, Double-Blinded, Randomized Controlled Trial Comparing the Efficacy of Adductor Canal Pain Catheters Following Total Knee Arthroplasty
Brief Title: A Study to Compare the Effectiveness of Adductor Canal Pain Catheters Following Total Knee Arthroplasty
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Benjamin K. Wilke, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 21-000974
Record Dates: First submitted 2021-09-13; First posted 2021-09-22 (Actual); Results first posted 2024-02-22 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: A Three-Arm, Double-Blinded, Randomized Controlled Trial
Who Masked: Participant, Investigator
Masking Description: This will be a double-blinded study. Computer randomization will be used for patient grouping and the research pharmacy will dispense the medication to the anesthesia team, who will set the adductor catheter dosing based upon randomization. The surgical team and patient will remain blinded to the medication and dosing regimen.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Ropivacaine intermittent bolus (Experimental): Subjects will have a catheter placed in the Post Anesthesia Care Unit following clinically indicated surgery with 0.2% ropivacaine dispersed in pulsed intermittent bolus.
  Interventions: Drug: Ropivacaine Intermittent Bolus
- Ropivacaine continuous (Experimental): Subjects will have a catheter placed in the Post Anesthesia Care Unit following clinically indicated surgery with 0.2% ropivacaine dispersed in a continuous infusion.
  Interventions: Drug: Ropivacaine Continuous Infusion
- Single shot adductor canal (Placebo Comparator): Subjects will have a catheter placed in the Post Anesthesia Care Unit following clinically indicated surgery with saline.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ropivacaine Continuous Infusion — 0.2% continuous infusion 6mL/hr
  Arms: Ropivacaine continuous
Drug: Ropivacaine Intermittent Bolus — 0.2% intermittent bolus infusion 8mL every 2 hours
  Arms: Ropivacaine intermittent bolus
Drug: Placebo — Saline filled catheter
  Arms: Single shot adductor canal

SUMMARY:
The purpose of this research is to study how well the adductor canal pain catheters works after a total knee arthroplasty or replacement of the knee joint. The catheter works by using either an intermittent bolus injection to provide a large dose of medication or continuous infusion of pain medicine, ropivacaine 0.2%, compared to a single-shot adductor canal block.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 and ≤ 90 years.
* Willing to participate in the study and competent to provide informed consent.
* Willing to comply with protocol procedures.
* Has an underlying diagnosis of osteoarthritis indicated for a total knee arthroplasty.

Exclusion Criteria:

* The patient must not have taken any narcotic medications (schedule II) during the 3 months leading up to the surgery.
* The patient must not be allergic or intolerant to a medication used in the multimodal pain pathway.
* Revision knee arthroplasty.
* Uncontrolled diabetes with A1C > 8.0%.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-04-13 (Actual); Primary Completion 2023-02-27 (Actual); Study Completion 2023-02-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Wilke, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Groups:
- Single Shot Adductor Canal: Subjects had a catheter placed in the Post Anesthesia Care Unit following clinically indicated surgery with saline.
  Placebo: Saline filled catheter
- Ropivacaine Continuous: Subjects had a catheter placed in the Post Anesthesia Care Unit following clinically indicated surgery with 0.2% ropivacaine dispersed in a continuous infusion.
  Ropivacaine Continuous Infusion: 0.2% continuous infusion 6mL/hr
- Ropivacaine Intermittent Bolus: Subjects had a catheter placed in the Post Anesthesia Care Unit following clinically indicated surgery with 0.2% ropivacaine dispersed in pulsed intermittent bolus.
  Ropivacaine Intermittent Bolus: 0.2% intermittent bolus infusion 8mL every 2 hours
Period: Overall Study
Arm/Group | Single Shot Adductor Canal | Ropivacaine Continuous | Ropivacaine Intermittent Bolus
Started | 21 | 20 | 19
Completed | 21 | 20 | 19
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Single Shot Adductor Canal | Ropivacaine Continuous | Ropivacaine Intermittent Bolus | Total
Number analyzed (Participants) | 21 | 20 | 19 | 60
Age, Continuous [Median (Full Range); unit: years] | 75 [52 to 81] | 71 [49 to 80] | 70 [52 to 79] | 72 [49 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 7 | 12 | 34
  Male | 6 | 13 | 7 | 26
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 18 | 19 | 18 | 55
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 3 | 1 | 1 | 5
Region of Enrollment [Number; unit: participants]
  United States | 21 | 20 | 19 | 60

OUTCOME MEASURES:

1. Primary Outcome: Post-operative Pain Levels
Description: Patient self-reported pain intensity score measured on the Visual Analogue Scale (VAS) rated from 0-10, where 0 was no pain and 10 was the worst pain imaginable.
Time Frame: 14 days post-operatively
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Single Shot Adductor Canal | Ropivacaine Continuous | Ropivacaine Intermittent Bolus
Number analyzed (Participants) | 21 | 20 | 19
score on a scale | 5.1 [1.7 to 7.9] | 5.1 [3.1 to 8.3] | 6.1 [1.9 to 8.0]

2. Secondary Outcome: Amount of Medication Administered
Description: Amount of medication administered via the patient-controlled function on the adductor catheter
Time Frame: 60 days, or until discontinuation of narcotic medication (whichever is later)
Measure: Median (Full Range); unit: mL
Arm/Group | Single Shot Adductor Canal | Ropivacaine Continuous | Ropivacaine Intermittent Bolus
Number analyzed (Participants) | 21 | 20 | 19
mL | 138 [18 to 222] | 111 [6 to 222] | 144 [24 to 240]

3. Secondary Outcome: Duration of Narcotic Used
Description: Number of days that narcotic use was required.
Time Frame: 60 days, or until discontinuation of narcotic medication (whichever is later)
Measure: Median (Full Range); unit: days
Arm/Group | Single Shot Adductor Canal | Ropivacaine Continuous | Ropivacaine Intermittent Bolus
Number analyzed (Participants) | 21 | 20 | 19
days | 21 [1 to 60] | 14 [5 to 60] | 14 [2 to 60]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from baseline to end of study, approximately, 60 days
Arm/Group | Single Shot Adductor Canal | Ropivacaine Continuous | Ropivacaine Intermittent Bolus
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/20 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/20 | 0/19
Other Adverse Events (participants affected / at risk) | 0/21 | 3/20 | 2/19
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Shot Adductor Canal (N=21) | Ropivacaine Continuous (N=20) | Ropivacaine Intermittent Bolus (N=19)
Catheter removed early (Surgical and medical procedures) | 0 (0) | 2 | 1
Catheter placed incorrectly (Surgical and medical procedures) | 0 | 0 | 1
Fever (General disorders) | 0 | 0 | 1
Knew swelling (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Knee bruising (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-12-13): https://cdn.clinicaltrials.gov/large-docs/87/NCT05053087/Prot_SAP_000.pdf